CLINICAL TRIAL: NCT05808101
Title: Role of the Gut Microbiome as Determinant of Depression in Multiple Sclerosis Subjects
Brief Title: Gut Microbiome and Depression
Status: Terminated | Type: Observational
Why Stopped: Change in PI and lack of personnel available to complete futher enrollment
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Connecticut (Other); University of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 202107067
Record Dates: First submitted 2022-05-17; First posted 2023-04-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis; Depression
Keywords: Multiple Sclerosis; Depression; Microbiome
MeSH Terms: conditions — Multiple Sclerosis; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A peripheral blood sample will be obtained from each participant to perform: 1) peripheral blood immune cell phenotyping to characterize the main immune cell subsets and their activation; 2) intracellular cytokine production to study cytokine production profiles of blood lymphocytes and monocytes.
  Stool samples will be processed for microbiome sequencing and metabolome characterization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Neuro-QoL Depression scale T-score > 55: 1. Collection of demographic and clinical data (age, gender, BMI, ethnicity, age of onset, number of relapses).
  2. Administration of the Neuro-QoL depression scale
  3. Neurological exam to evaluate disability and calculate the EDSS score (ranging from 0 to 10)
  4. Neurological cognitive and functional assessments: a 9-hole Peg Test and 25-ft Timed Walk from the Multiple Sclerosis Functional Composite (MSFC); the Symbol Digit Modality Test (SDMT)
  5. Administration of the Fatigue Severity Scale (FSS)
  6. Collection of a 4-days food diary to evaluate diet composition of enrolled pwMS
  7. Administration of the Stanford 7-day Physical Activity Recall Scale (PAR)
  8. Evaluation of sleep quality by administration of the Neuro-QoL sleep disturbance scale
  9. Collection of a stool sample for gut microbiome and metabolome analyses
  10. Collection of a saliva sample for microbiome and metabolome analyses
  Interventions: Other: Neuro-QoL T-score determination
- With Neuro-QoL Depression scale T-score < 55: 1. Collection of demographic and clinical data (age, gender, BMI, ethnicity, age of onset, number of relapses).
  2. Administration of the Neuro-QoL depression scale
  3. Neurological exam to evaluate disability and calculate the EDSS score (ranging from 0 to 10)
  4. Neurological cognitive and functional assessments: a 9-hole Peg Test and 25-ft Timed Walk from the Multiple Sclerosis Functional Composite (MSFC); the Symbol Digit Modality Test (SDMT)
  5. Administration of the Fatigue Severity Scale (FSS)
  6. Collection of a 4-days food diary to evaluate diet composition of enrolled pwMS
  7. Administration of the Stanford 7-day Physical Activity Recall Scale (PAR)
  8. Evaluation of sleep quality by administration of the Neuro-QoL sleep disturbance scale
  9. Collection of a stool sample for gut microbiome and metabolome analyses
  10. Collection of a saliva sample for microbiome and metabolome analyses
  Interventions: Other: Neuro-QoL T-score determination

INTERVENTIONS:
Other: Neuro-QoL T-score determination — Neuro-Qol depression scale, using a T-score of 55 as a threshold

SUMMARY:
The purpose of this project is to determine if specific gut microbiome or gut-derived metabolites are associated with depression in patients with Multiple Sclerosis (pwMS). Mechanistically, the investigators further hypothesize that depression in pwMS is related to decreased abundance of gut bacteria with GABA-producing activities and/or with anti-inflammatory properties. To determine if the presence of depression in pwMS is associated with specific gut microbiome, gut-derived metabolites or peripheral blood immune profiles. The investigators will perform a cross-sectional study in clinically stable pwMS recruited at the John L. Trotter MS Center. The investigators will evaluate the presence of depression using the Quality of Life in Neurological Disorders (Neuro-Qol) depression scale, one of the 13 scales in the Neuro-Qol recently developed by the NIH using modern psychometric techniques and validated in pwMS.

A total of 120 pwMS will be recruited: 60 with and 60 without depression based on the Neuro-Qol depression scale. At the study visit each participant will be asked to provide a stool sample for microbiome analyses and a blood sample for peripheral blood immunophenotyping. Potential confounders will be collected and treated as covariates in the analyses. These include: 1) degree of disability (EDSS); 2) treatment with anti-depressants and DMTs; 3) a 4-days food diary to evaluate diet composition; 4) weight and height to calculate the BMI; 5) fatigue; 6) level of physical activity; 7) sleep quality.

DETAILED DESCRIPTION:
Our overall hypothesis is that specific gut microbiome or gut-derived metabolites are associated with depression in pwMS. Mechanistically, the investigators further hypothesize that depression in pwMS is related to decreased abundance of gut bacteria with GABA-producing activities and/or with anti-inflammatory properties.

AIM 1. To determine if the presence of depression in pwMS is associated with specific gut microbiome, gut-derived metabolites or peripheral blood immune profiles.

The investigators will perform a cross-sectional study in clinically stable pwMS recruited at the John L. Trotter MS Center. The investigators will evaluate the presence of depression using the Quality of Life in Neurological Disorders (Neuro-Qol) depression scale, one of the 13 scales in the Neuro-Qol recently developed by the NIH using modern psychometric techniques and validated in pwMS. A total of 120 pwMS will be recruited: 60 with and 60 without depression based on the Neuro-Qol depression scale. At the study visit each participant will be asked to provide a stool sample for microbiome analyses and a blood sample for peripheral blood immunophenotyping. Potential confounders will be collected and treated as covariates in the analyses. These include: 1) degree of disability (EDSS); 2) treatment with anti-depressants and DMTs; 3) a 4-days food diary to evaluate diet composition; 4) the investigatorsight and height to calculate the BMI; 5) fatigue; 6) level of physical activity; 7) sleep quality.

AIM 1A. To determine if depression will correlate with specific gut microbiome or gut-derived metabolites profiles in pwMS.

Stool samples will be processed for microbiome sequencing and metabolome characterization.

AIM 1B. To determine if depression will correlate with a specific peripheral blood immune-inflammatory profile in pwMS.

A peripheral blood sample will be obtained from each participant to perform: 1) peripheral blood immune cell phenotyping to characterize the main immune cell subsets and their activation; 2) intracellular cytokine production to study cytokine production profiles of blood lymphocytes and monocytes.

AIM 2. To quantify GABA production in pwMS with or without depression and determine gut microbiome-immune system interaction in vitro.

In this aim the investigators will perform functional studies to evaluate the potential of gut microbiota from pwMS with or without depression to produce GABA and to modulate immune-inflammatory responses.

AIM 2A. To quantify GABA levels in whole stool, specific stool bacterial isolates and blood of pwMS with or without depression.

The investigators will evaluate GABA levels in the stool and blood of pwMS. In addition, the investigators will measure GABA production by Bacteroides ssp isolated from the gut microbiota of pwMS.

Aim 2B. To evaluate the effects of whole stool and specific bacterial species from pwMS on blood immune cell phenotype and cytokine production.

The investigators will test how whole gut microbiome or specific bacteria (identified in Aim 1 as associated with depression in pwMS) can modulate immune cell function. Peripheral blood mononuclear cells (PBMC) from healthy donors will be cultured in conditioning media from whole stool or bacteria of interest isolated from pwMS. PBMC phenotype and cytokine production after exposure in vitro will be characterized by flow cytometry.

ELIGIBILITY:
1. Age ≥18 years
2. Diagnosis of RRMS or progressive MS based on the 2017 revised McDonald criteria
3. Untreated or on any of the MS DMTs as long as they have been stable clinically in the previous 3 months
4. No history of antibiotic treatment in the 3 months prior to study visit and sample collection
5. No other autoimmune diseases, chronic metabolic diseases (e.g. diabetes) or conditions (e.g. pregnancy) that would interfere with the parameters that we will be measuring in the stool and blood samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis (MS)
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Gut microbiome, gut-derived metabolites and peripheral blood immune profiles | 3 years
  Gut microbiome will be characterized by metagenomic sequencing. Untargeted metabolome analysis performed by LC-MS. Peripheral blood phenotyping performed by flow cytometry analysis
GABA levels in whole stool, specific stool bacteria isolates and blood | 3 Years
  GABA levels in whole stool measured by targeted LC-MS Effects of whole stool and specific bacterial species from people with MS with or without depression on blood immune cell phenotype and cytokine production measured by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Piccio, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will be determined based whether or not recruitment numbers will be sufficient to power outcome analyses.

REFERENCES:
- [Background] Feinstein A, Magalhaes S, Richard JF, Audet B, Moore C. The link between multiple sclerosis and depression. Nat Rev Neurol. 2014 Sep;10(9):507-17. doi: 10.1038/nrneurol.2014.139. Epub 2014 Aug 12. PMID 25112509
- [Background] Liu Y, Tang X. Depressive Syndromes in Autoimmune Disorders of the Nervous System: Prevalence, Etiology, and Influence. Front Psychiatry. 2018 Sep 25;9:451. doi: 10.3389/fpsyt.2018.00451. eCollection 2018. PMID 30319458
- [Background] Flux MC, Lowry CA. Finding intestinal fortitude: Integrating the microbiome into a holistic view of depression mechanisms, treatment, and resilience. Neurobiol Dis. 2020 Feb;135:104578. doi: 10.1016/j.nbd.2019.104578. Epub 2019 Aug 24. PMID 31454550
- [Background] Zheng P, Zeng B, Zhou C, Liu M, Fang Z, Xu X, Zeng L, Chen J, Fan S, Du X, Zhang X, Yang D, Yang Y, Meng H, Li W, Melgiri ND, Licinio J, Wei H, Xie P. Gut microbiome remodeling induces depressive-like behaviors through a pathway mediated by the host's metabolism. Mol Psychiatry. 2016 Jun;21(6):786-96. doi: 10.1038/mp.2016.44. Epub 2016 Apr 12. PMID 27067014
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Wallace CJK, Milev R. The effects of probiotics on depressive symptoms in humans: a systematic review. Ann Gen Psychiatry. 2017 Feb 20;16:14. doi: 10.1186/s12991-017-0138-2. eCollection 2017. PMID 28239408
- [Background] Valles-Colomer M, Falony G, Darzi Y, Tigchelaar EF, Wang J, Tito RY, Schiweck C, Kurilshikov A, Joossens M, Wijmenga C, Claes S, Van Oudenhove L, Zhernakova A, Vieira-Silva S, Raes J. The neuroactive potential of the human gut microbiota in quality of life and depression. Nat Microbiol. 2019 Apr;4(4):623-632. doi: 10.1038/s41564-018-0337-x. Epub 2019 Feb 4. PMID 30718848
- [Background] Dethloff F, Vargas F, Elijah E, Quinn R, Park DI, Herzog DP, Muller MB, Gentry EC, Knight R, Gonzalez A, Dorrestein PC, Turck CW. Paroxetine Administration Affects Microbiota and Bile Acid Levels in Mice. Front Psychiatry. 2020 Jun 4;11:518. doi: 10.3389/fpsyt.2020.00518. eCollection 2020. PMID 32581888
- [Background] McGovern AS, Hamlin AS, Winter G. A review of the antimicrobial side of antidepressants and its putative implications on the gut microbiome. Aust N Z J Psychiatry. 2019 Dec;53(12):1151-1166. doi: 10.1177/0004867419877954. Epub 2019 Sep 26. PMID 31558039
- [Background] van den Hoogen WJ, Laman JD, 't Hart BA. Modulation of Multiple Sclerosis and Its Animal Model Experimental Autoimmune Encephalomyelitis by Food and Gut Microbiota. Front Immunol. 2017 Sep 5;8:1081. doi: 10.3389/fimmu.2017.01081. eCollection 2017. PMID 28928747
- [Background] Cantarel BL, Waubant E, Chehoud C, Kuczynski J, DeSantis TZ, Warrington J, Venkatesan A, Fraser CM, Mowry EM. Gut microbiota in multiple sclerosis: possible influence of immunomodulators. J Investig Med. 2015 Jun;63(5):729-34. doi: 10.1097/JIM.0000000000000192. PMID 25775034
- [Background] Berer K, Gerdes LA, Cekanaviciute E, Jia X, Xiao L, Xia Z, Liu C, Klotz L, Stauffer U, Baranzini SE, Kumpfel T, Hohlfeld R, Krishnamoorthy G, Wekerle H. Gut microbiota from multiple sclerosis patients enables spontaneous autoimmune encephalomyelitis in mice. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10719-10724. doi: 10.1073/pnas.1711233114. Epub 2017 Sep 11. PMID 28893994
- [Background] Cekanaviciute E, Yoo BB, Runia TF, Debelius JW, Singh S, Nelson CA, Kanner R, Bencosme Y, Lee YK, Hauser SL, Crabtree-Hartman E, Sand IK, Gacias M, Zhu Y, Casaccia P, Cree BAC, Knight R, Mazmanian SK, Baranzini SE. Gut bacteria from multiple sclerosis patients modulate human T cells and exacerbate symptoms in mouse models. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10713-10718. doi: 10.1073/pnas.1711235114. Epub 2017 Sep 11. PMID 28893978
- [Background] Jangi S, Gandhi R, Cox LM, Li N, von Glehn F, Yan R, Patel B, Mazzola MA, Liu S, Glanz BL, Cook S, Tankou S, Stuart F, Melo K, Nejad P, Smith K, Topcuolu BD, Holden J, Kivisakk P, Chitnis T, De Jager PL, Quintana FJ, Gerber GK, Bry L, Weiner HL. Alterations of the human gut microbiome in multiple sclerosis. Nat Commun. 2016 Jun 28;7:12015. doi: 10.1038/ncomms12015. PMID 27352007
- [Background] Dinan TG, Cryan JF. Gut instincts: microbiota as a key regulator of brain development, ageing and neurodegeneration. J Physiol. 2017 Jan 15;595(2):489-503. doi: 10.1113/JP273106. Epub 2016 Dec 4. PMID 27641441
- [Background] Kim YK, Na KS, Shin KH, Jung HY, Choi SH, Kim JB. Cytokine imbalance in the pathophysiology of major depressive disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jun 30;31(5):1044-53. doi: 10.1016/j.pnpbp.2007.03.004. Epub 2007 Mar 13. PMID 17433516
- [Background] Kelly JR, Kennedy PJ, Cryan JF, Dinan TG, Clarke G, Hyland NP. Breaking down the barriers: the gut microbiome, intestinal permeability and stress-related psychiatric disorders. Front Cell Neurosci. 2015 Oct 14;9:392. doi: 10.3389/fncel.2015.00392. eCollection 2015. PMID 26528128
- [Background] Braniste V, Al-Asmakh M, Kowal C, Anuar F, Abbaspour A, Toth M, Korecka A, Bakocevic N, Ng LG, Kundu P, Gulyas B, Halldin C, Hultenby K, Nilsson H, Hebert H, Volpe BT, Diamond B, Pettersson S. The gut microbiota influences blood-brain barrier permeability in mice. Sci Transl Med. 2014 Nov 19;6(263):263ra158. doi: 10.1126/scitranslmed.3009759. PMID 25411471
- [Background] Parada Venegas D, De la Fuente MK, Landskron G, Gonzalez MJ, Quera R, Dijkstra G, Harmsen HJM, Faber KN, Hermoso MA. Corrigendum: Short Chain Fatty Acids (SCFAs)-Mediated Gut Epithelial and Immune Regulation and Its Relevance for Inflammatory Bowel Diseases. Front Immunol. 2019 Jun 28;10:1486. doi: 10.3389/fimmu.2019.01486. eCollection 2019. PMID 31316522
- [Background] Strandwitz P. Neurotransmitter modulation by the gut microbiota. Brain Res. 2018 Aug 15;1693(Pt B):128-133. doi: 10.1016/j.brainres.2018.03.015. PMID 29903615
- [Background] Yano JM, Yu K, Donaldson GP, Shastri GG, Ann P, Ma L, Nagler CR, Ismagilov RF, Mazmanian SK, Hsiao EY. Indigenous bacteria from the gut microbiota regulate host serotonin biosynthesis. Cell. 2015 Apr 9;161(2):264-76. doi: 10.1016/j.cell.2015.02.047. Erratum In: Cell. 2015 Sep 24;163:258. PMID 25860609
- [Background] Fogaca MV, Duman RS. Cortical GABAergic Dysfunction in Stress and Depression: New Insights for Therapeutic Interventions. Front Cell Neurosci. 2019 Mar 12;13:87. doi: 10.3389/fncel.2019.00087. eCollection 2019. PMID 30914923
- [Background] Kalueff AV, Nutt DJ. Role of GABA in anxiety and depression. Depress Anxiety. 2007;24(7):495-517. doi: 10.1002/da.20262. PMID 17117412
- [Background] Pehrson AL, Sanchez C. Altered gamma-aminobutyric acid neurotransmission in major depressive disorder: a critical review of the supporting evidence and the influence of serotonergic antidepressants. Drug Des Devel Ther. 2015 Jan 19;9:603-24. doi: 10.2147/DDDT.S62912. eCollection 2015. PMID 25653499
- [Background] Strandwitz P, Kim KH, Terekhova D, Liu JK, Sharma A, Levering J, McDonald D, Dietrich D, Ramadhar TR, Lekbua A, Mroue N, Liston C, Stewart EJ, Dubin MJ, Zengler K, Knight R, Gilbert JA, Clardy J, Lewis K. GABA-modulating bacteria of the human gut microbiota. Nat Microbiol. 2019 Mar;4(3):396-403. doi: 10.1038/s41564-018-0307-3. Epub 2018 Dec 10. PMID 30531975
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Minden SL, Feinstein A, Kalb RC, Miller D, Mohr DC, Patten SB, Bever C Jr, Schiffer RB, Gronseth GS, Narayanaswami P; Guideline Development Subcommittee of the American Academy of Neurology. Evidence-based guideline: assessment and management of psychiatric disorders in individuals with MS: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2014 Jan 14;82(2):174-81. doi: 10.1212/WNL.0000000000000013. Epub 2013 Dec 27. PMID 24376275
- [Background] Lee CH, Giuliani F. The Role of Inflammation in Depression and Fatigue. Front Immunol. 2019 Jul 19;10:1696. doi: 10.3389/fimmu.2019.01696. eCollection 2019. PMID 31379879
- [Background] Sharon G, Sampson TR, Geschwind DH, Mazmanian SK. The Central Nervous System and the Gut Microbiome. Cell. 2016 Nov 3;167(4):915-932. doi: 10.1016/j.cell.2016.10.027. PMID 27814521
- [Background] Sokol H, Pigneur B, Watterlot L, Lakhdari O, Bermudez-Humaran LG, Gratadoux JJ, Blugeon S, Bridonneau C, Furet JP, Corthier G, Grangette C, Vasquez N, Pochart P, Trugnan G, Thomas G, Blottiere HM, Dore J, Marteau P, Seksik P, Langella P. Faecalibacterium prausnitzii is an anti-inflammatory commensal bacterium identified by gut microbiota analysis of Crohn disease patients. Proc Natl Acad Sci U S A. 2008 Oct 28;105(43):16731-6. doi: 10.1073/pnas.0804812105. Epub 2008 Oct 20. PMID 18936492
- [Background] Depommier C, Everard A, Druart C, Plovier H, Van Hul M, Vieira-Silva S, Falony G, Raes J, Maiter D, Delzenne NM, de Barsy M, Loumaye A, Hermans MP, Thissen JP, de Vos WM, Cani PD. Supplementation with Akkermansia muciniphila in overweight and obese human volunteers: a proof-of-concept exploratory study. Nat Med. 2019 Jul;25(7):1096-1103. doi: 10.1038/s41591-019-0495-2. Epub 2019 Jul 1. PMID 31263284
- [Background] Bhat R, Axtell R, Mitra A, Miranda M, Lock C, Tsien RW, Steinman L. Inhibitory role for GABA in autoimmune inflammation. Proc Natl Acad Sci U S A. 2010 Feb 9;107(6):2580-5. doi: 10.1073/pnas.0915139107. Epub 2010 Feb 1. PMID 20133656
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Sandoval-Salazar C, Ramirez-Emiliano J, Trejo-Bahena A, Oviedo-Solis CI, Solis-Ortiz MS. A high-fat diet decreases GABA concentration in the frontal cortex and hippocampus of rats. Biol Res. 2016 Feb 29;49:15. doi: 10.1186/s40659-016-0075-6. PMID 26927389
- [Background] Belkaid Y, Hand TW. Role of the microbiota in immunity and inflammation. Cell. 2014 Mar 27;157(1):121-41. doi: 10.1016/j.cell.2014.03.011. PMID 24679531
- [Background] Lassmann H, Bradl M. Multiple sclerosis: experimental models and reality. Acta Neuropathol. 2017 Feb;133(2):223-244. doi: 10.1007/s00401-016-1631-4. Epub 2016 Oct 20. PMID 27766432
- [Background] Hausser-Kinzel S, Weber MS. The Role of B Cells and Antibodies in Multiple Sclerosis, Neuromyelitis Optica, and Related Disorders. Front Immunol. 2019 Feb 8;10:201. doi: 10.3389/fimmu.2019.00201. eCollection 2019. PMID 30800132
- [Background] Ahmetspahic D, Schwarte K, Ambree O, Burger C, Falcone V, Seiler K, Kooybaran MR, Grosse L, Roos F, Scheffer J, Jorgens S, Koelkebeck K, Dannlowski U, Arolt V, Scheu S, Alferink J. Altered B Cell Homeostasis in Patients with Major Depressive Disorder and Normalization of CD5 Surface Expression on Regulatory B Cells in Treatment Responders. J Neuroimmune Pharmacol. 2018 Mar;13(1):90-99. doi: 10.1007/s11481-017-9763-4. Epub 2017 Sep 13. PMID 28905187
- [Background] Miller DM, Bethoux F, Victorson D, Nowinski CJ, Buono S, Lai JS, Wortman K, Burns JL, Moy C, Cella D. Validating Neuro-QoL short forms and targeted scales with people who have multiple sclerosis. Mult Scler. 2016 May;22(6):830-41. doi: 10.1177/1352458515599450. Epub 2015 Aug 3. PMID 26238464
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Mowry EM, Bermel RA, Williams JR, Benzinger TLS, de Moor C, Fisher E, Hersh CM, Hyland MH, Izbudak I, Jones SE, Kieseier BC, Kitzler HH, Krupp L, Lui YW, Montalban X, Naismith RT, Nicholas JA, Pellegrini F, Rovira A, Schulze M, Tackenberg B, Tintore M, Tivarus ME, Ziemssen T, Rudick RA. Harnessing Real-World Data to Inform Decision-Making: Multiple Sclerosis Partners Advancing Technology and Health Solutions (MS PATHS). Front Neurol. 2020 Aug 7;11:632. doi: 10.3389/fneur.2020.00632. eCollection 2020. PMID 32849170
- [Background] Guenther PM, Casavale KO, Reedy J, Kirkpatrick SI, Hiza HA, Kuczynski KJ, Kahle LL, Krebs-Smith SM. Update of the Healthy Eating Index: HEI-2010. J Acad Nutr Diet. 2013 Apr;113(4):569-80. doi: 10.1016/j.jand.2012.12.016. Epub 2013 Feb 13. PMID 23415502
- [Background] Sallis JF, Haskell WL, Wood PD, Fortmann SP, Rogers T, Blair SN, Paffenbarger RS Jr. Physical activity assessment methodology in the Five-City Project. Am J Epidemiol. 1985 Jan;121(1):91-106. doi: 10.1093/oxfordjournals.aje.a113987. PMID 3964995
- [Background] Zhou W, Sailani MR, Contrepois K, Zhou Y, Ahadi S, Leopold SR, Zhang MJ, Rao V, Avina M, Mishra T, Johnson J, Lee-McMullen B, Chen S, Metwally AA, Tran TDB, Nguyen H, Zhou X, Albright B, Hong BY, Petersen L, Bautista E, Hanson B, Chen L, Spakowicz D, Bahmani A, Salins D, Leopold B, Ashland M, Dagan-Rosenfeld O, Rego S, Limcaoco P, Colbert E, Allister C, Perelman D, Craig C, Wei E, Chaib H, Hornburg D, Dunn J, Liang L, Rose SMS, Kukurba K, Piening B, Rost H, Tse D, McLaughlin T, Sodergren E, Weinstock GM, Snyder M. Longitudinal multi-omics of host-microbe dynamics in prediabetes. Nature. 2019 May;569(7758):663-671. doi: 10.1038/s41586-019-1236-x. Epub 2019 May 29. PMID 31142858
- [Background] Smith CA, Want EJ, O'Maille G, Abagyan R, Siuzdak G. XCMS: processing mass spectrometry data for metabolite profiling using nonlinear peak alignment, matching, and identification. Anal Chem. 2006 Feb 1;78(3):779-87. doi: 10.1021/ac051437y. PMID 16448051
- [Background] Chong J, Soufan O, Li C, Caraus I, Li S, Bourque G, Wishart DS, Xia J. MetaboAnalyst 4.0: towards more transparent and integrative metabolomics analysis. Nucleic Acids Res. 2018 Jul 2;46(W1):W486-W494. doi: 10.1093/nar/gky310. PMID 29762782
- [Background] Longbrake EE, Ramsbottom MJ, Cantoni C, Ghezzi L, Cross AH, Piccio L. Dimethyl fumarate selectively reduces memory T cells in multiple sclerosis patients. Mult Scler. 2016 Jul;22(8):1061-1070. doi: 10.1177/1352458515608961. Epub 2015 Oct 12. PMID 26459150
- [Background] Ghezzi L, Cantoni C, Cignarella F, Bollman B, Cross AH, Salter A, Galimberti D, Cella M, Piccio L. T cells producing GM-CSF and IL-13 are enriched in the cerebrospinal fluid of relapsing MS patients. Mult Scler. 2020 Sep;26(10):1172-1186. doi: 10.1177/1352458519852092. Epub 2019 Jun 25. PMID 31237799
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biol Psychiatry. 2009 May 1;65(9):732-41. doi: 10.1016/j.biopsych.2008.11.029. Epub 2009 Jan 15. PMID 19150053
- [Background] Luscher B, Shen Q, Sahir N. The GABAergic deficit hypothesis of major depressive disorder. Mol Psychiatry. 2011 Apr;16(4):383-406. doi: 10.1038/mp.2010.120. Epub 2010 Nov 16. PMID 21079608
- [Background] Auteri M, Zizzo MG, Serio R. GABA and GABA receptors in the gastrointestinal tract: from motility to inflammation. Pharmacol Res. 2015 Mar;93:11-21. doi: 10.1016/j.phrs.2014.12.001. Epub 2014 Dec 17. PMID 25526825
- [Background] Fujimura KE, Sitarik AR, Havstad S, Lin DL, Levan S, Fadrosh D, Panzer AR, LaMere B, Rackaityte E, Lukacs NW, Wegienka G, Boushey HA, Ownby DR, Zoratti EM, Levin AM, Johnson CC, Lynch SV. Neonatal gut microbiota associates with childhood multisensitized atopy and T cell differentiation. Nat Med. 2016 Oct;22(10):1187-1191. doi: 10.1038/nm.4176. Epub 2016 Sep 12. PMID 27618652
- [Background] Dhakal R, Bajpai VK, Baek KH. Production of gaba (gamma - Aminobutyric acid) by microorganisms: a review. Braz J Microbiol. 2012 Oct;43(4):1230-41. doi: 10.1590/S1517-83822012000400001. Epub 2012 Jun 1. PMID 24031948
- [Background] Pokusaeva K, Johnson C, Luk B, Uribe G, Fu Y, Oezguen N, Matsunami RK, Lugo M, Major A, Mori-Akiyama Y, Hollister EB, Dann SM, Shi XZ, Engler DA, Savidge T, Versalovic J. GABA-producing Bifidobacterium dentium modulates visceral sensitivity in the intestine. Neurogastroenterol Motil. 2017 Jan;29(1):e12904. doi: 10.1111/nmo.12904. Epub 2016 Jul 25. PMID 27458085
- [Background] Cuypers K, Maes C, Swinnen SP. Aging and GABA. Aging (Albany NY). 2018 Jun 13;10(6):1186-1187. doi: 10.18632/aging.101480. No abstract available. PMID 29905530
- [Background] Boonstra E, de Kleijn R, Colzato LS, Alkemade A, Forstmann BU, Nieuwenhuis S. Neurotransmitters as food supplements: the effects of GABA on brain and behavior. Front Psychol. 2015 Oct 6;6:1520. doi: 10.3389/fpsyg.2015.01520. eCollection 2015. PMID 26500584
- [Background] Schirmer M, Smeekens SP, Vlamakis H, Jaeger M, Oosting M, Franzosa EA, Horst RT, Jansen T, Jacobs L, Bonder MJ, Kurilshikov A, Fu J, Joosten LAB, Zhernakova A, Huttenhower C, Wijmenga C, Netea MG, Xavier RJ. Linking the Human Gut Microbiome to Inflammatory Cytokine Production Capacity. Cell. 2016 Dec 15;167(7):1897. doi: 10.1016/j.cell.2016.11.046. No abstract available. PMID 27984736